CLINICAL TRIAL: NCT00453557
Title: Mechanism of Growth Hormone Effects on Adipose Tissue
Acronym: GH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Frank Greenway, Clinical Medical Doctor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 99009
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Obesity
Keywords: growth hormone, obesity, visceral adiposity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: rhGH

SUMMARY:
Growth hormone treatment in humans has been shown to decrease body fat. This study aims to determine what adipose tissue depots are affected by GH and what is the mechanism.

DETAILED DESCRIPTION:
Growth hormone (GH) replacement in GH deficient adults results in an improvement in metabolic status, an increase in lean body mass and a reduction in visceral adiposity. GH might also decrease visceral adiposity in obese adults that are not GH deficient.

The objective of the study is to determine the effects of GH on the metabolic syndrome and visceral adiposity in men with low blood levels of IGF-1 and the durability of these effects after stopping GH therapy. We will use a double blind, placebo controlled 6 month intervention trial followed by a blinded follow-up period of 6 months. Thirty non-diabetic middle aged men with central adiposity (BMI > 27 kg/m2, waist circumference > 102 cm) will participate.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 40-70
* Central obesity defined as waist circumference greater than 102 cm and BMI > 27 and < 35 kg/m2
* No weight loss in last 12 months
* Total IGF-1 level < 241 ng/ml (~25th percentile for the assay)
* Body habitus which permitted accurate CT scan acquisition and analysis.

Exclusion Criteria:

* Significant neurologic, metabolic, endocrine, cardiac, respiratory or gastrointestinal disease
* Diabetes
* Known coronary heart disease
* Exercised more than 3 hours per week
* Unwilling or unable to abstain from alcohol for 72 hours prior to the measurements of energy expenditure and fasting blood work

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 1999-04; Primary Completion 2000-12 (Actual); Study Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
body composition at baseline, after 6 months of treatment and at the end of the followup period
energy expenditure at baseline, after 6 months of treatment and at the end of the followup period

SECONDARY OUTCOMES:
gene expression in adipose tissue at baseline and after 6 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Smith, M.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States